CLINICAL TRIAL: NCT04724603
Title: Phage Safety Retrospective Cohort Study
Acronym: PHASACO-retro
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 334
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-09

CONDITIONS: Bone and Joint Infection; Prosthetic Joint Infection
Keywords: bone and joint infection; phagotherapy; adverse event; Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having had avderse event after phagotherapy for bone or joint infection
  Interventions: Other: patients having had avderse event after phagotherapy for bone or joint or implant infection

INTERVENTIONS:
Other: patients having had avderse event after phagotherapy for bone or joint or implant infection — to determine the accountability of adverse effects in having had avderse event after phagotherapy for bone or joint or implant infection

SUMMARY:
The aim of this study is to determine the imputability of adverse events in patients who have had phage therapy for the treatment of their bone or joint or implant infection, in order to find out whether these adverse effects are related to surgery, antibiotic treatment or bacteriophages.

ELIGIBILITY:
Inclusion Criteria:

* patients having had a bone or joint or implant infection treated by phagotherapy and having had an adverse event

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients having had a bone or joint or implant infection treated by phagotherapy at the CRIOAc Lyon and having had an adverse event
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
rate of patients having had an adverse event | 1 year
  number of patients having had an adverse event
rate of adverse event attributable to the surgery | 1 year
  number of patients having had an adverse event because of the surgery
type of adverse event attributable to the surgery | 1 year
  classification according to Clavien's Clasification
rate of adverse event attributable to the antibiotic treatment | 1 year
  number of patients having had an adverse event because of the antibiotic treatment
rate of adverse event attributable to the phagotherapy | 1 year
  number of patients having had an adverse event because of phagotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/